CLINICAL TRIAL: NCT04278898
Title: Targeting the Neurobiology of Restricted and Repetitive Behaviors in Children With Autism Using N-acetylcysteine: a Single-dose Challenge Study
Brief Title: Targeting the Neurobiology of RRB in Autism Using N-acetylcysteine: Single-dose
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Patrick Hegarty, Instructor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-54931; 1K99HD101702 (NIH)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Magnetic Resonance Imaging; N-acetylcysteine; Restricted and Repetitive Behaviors; electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine then Placebo (Experimental)
  Interventions: Drug: N-Acetylcysteine
- Placebo then N-acetylcysteine (Experimental)
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — N-acetylcysteine Single Dose 2700 mg taken orally

SUMMARY:
The goal of this study is to target the neurobiology of restricted and repetitive behaviors in children with autism spectrum disorder using N-acetylcysteine (NAC), a well-tolerated nutritional supplement that has shown promise for reducing symptom severity in recent small-scale trials. The findings from this research will shed light on the mechanisms of action underlying the clinical benefits of NAC.

ELIGIBILITY:
Inclusion Criteria:

* children between 3 years and 12 years 11 months at the time of consent
* diagnosis of Autism Spectrum Disorder confirmed with the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule-2 (ADOS-2), or Brief Observation of Symptoms of Autism (BOSA), or Childhood Autism Rating Scale- Second Edition (CARS-2).
* at least moderate Restricted and Repetitive Behaviors severity defined by a Children's Yale-Brown Obsessive Compulsive Scale for children with autism spectrum disorder score ≥ 11,
* physical development indicative of prepubescence as defined by the criteria for Tanner Stage 1,
* medically stable,
* passes MR safety screening (e.g., no metal in the body).

Exclusion Criteria:

* presence of known genetic abnormalities associated with Autism Spectrum Disorder (e.g. Fragile X),
* current or life-time diagnosis of severe psychiatric disorder (e.g., schizophrenia),
* presence of significant medical problems that would interfere with participation,
* the inability of at least one caregiver to speak/read English to a sufficient level to complete study requirements and materials,
* individuals taking antioxidant agents and glutathione prodrugs, or
* the inability/unwillingness to swallow an agent during the screening visit.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in glutamatergic neurometabolites (Glx) measured by proton spectroscopy Magnetic Resonance Imaging (MRI) | 1 hour after single dose

SECONDARY OUTCOMES:
Change in Gamma band amplitude and synchronization measured by electroencephalography | 1 hour after single dose

CONTACTS AND LOCATIONS:
Overall Officials: John Hegarty, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data will be shared with the National Database for Autism Research (NDAR)
Time Frame: The data will be submitted on January 15th and July 15th each year.
Access Criteria: Researchers with access to the National Database for Autism Research (NDAR) will be able to obtain the submitted data.
URL: https://nda.nih.gov/contribute/sharing-regimen.html